CLINICAL TRIAL: NCT07143708
Title: Comparison of the Safety and Efficacy of PreserFlo MicroShunt and XEN Stent Alone Versus With Amniotic Membrane in Glaucoma Surgery
Brief Title: Safety and Effectiveness of PreserFlo and XEN Stents With or Without Amniotic Membrane in Glaucoma Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Lesya Shuba, Principal Investigator, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1031327
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Glaucoma
Keywords: Galucoma; Glaucoma Surgery; Stent surgery; MicroShunt surgery
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Amniotic Membrane Group (Active Comparator): Patients receive standard glaucoma surgery (PreserFlo MicroShunt or XEN Stent) without additional covering. The choice between PreserFlo or XEN is not part of the study design-it's determined beforehand by the surgeon as part of regular care.
  Interventions: Other: Glaucoma Surgery without Amniotic Membrane
- Amniotic Membrane Group (Experimental): Patients receive standard glaucoma surgery (PreserFlo MicroShunt or XEN Stent) with additional covering. The implanted MicroShunt or Stent is covered with an amniotic membrane patch. The choice between PreserFlo or XEN is not part of the study design-it's determined beforehand by the surgeon as part of regular care.
  Interventions: Other: Glaucoma Surgery with Amniotic Membrane

INTERVENTIONS:
Other: Glaucoma Surgery with Amniotic Membrane — Arm 2: Glaucoma Surgery with Amniotic Membrane Participants undergo glaucoma surgery with either a PreserFlo MicroShunt or a XEN Stent, as determined by the treating surgeon. In this group, the implanted stent is covered with an amniotic membrane patch to reduce postoperative scarring and improve long-term outcomes. Follow-up visits are scheduled as per standard of care for glaucoma surgery (up to 12 months).
  Arms: Amniotic Membrane Group
Other: Glaucoma Surgery without Amniotic Membrane — Arm 1: Glaucoma Surgery without Amniotic Membrane Participants undergo glaucoma surgery with either a PreserFlo MicroShunt or a XEN Stent, as determined by the treating surgeon. No modifications are made to the procedure. Follow-up visits are scheduled as per standard of care for glaucoma surgery (up to 12 months).
  Arms: No Amniotic Membrane Group

SUMMARY:
Glaucoma is one of the leading causes of permanent blindness in the world. It happens when the optic nerve-the connection between the eye and the brain-is damaged. As this damage gets worse, vision is slowly lost.

Glaucoma treatments often begin with eye drops to lower eye pressure. If drops are not enough, surgery may be needed. The type of surgery depends on how advanced the glaucoma is and how much vision has already been lost.

Some glaucoma surgeries, including trabeculectomy, PreserFlo MicroShunt, and XEN Stent, create a new pathway for fluid to drain out of the eye. This helps lower pressure inside the eye.

However, after surgery, the body's natural healing process can sometimes cause inflammation and scarring, which may block the new drainage pathway. If this happens, eye pressure can rise again, and the surgery may not work as well as hoped.

This study is testing whether covering the PreserFlo or XEN devices with amniotic membrane (a safe tissue already used in other eye surgeries) can reduce scarring, improve healing, and lead to better long-term results. Amniotic membrane has already been used safely in many types of eye surgeries. It has been shown to improve healing and reduce scarring in some glaucoma surgeries. But it has not yet been studied in PreserFlo MicroShunt or XEN Stent procedures. The goal is to see if adding amniotic membrane makes the surgery safer and more effective for people with glaucoma.

DETAILED DESCRIPTION:
Glaucoma is the leading cause of permanent blindness worldwide. Glaucoma is damage to the optic nerve, which sends information from the eye to the brain. This damage causes vision to weaken. Treatment for glaucoma includes the use of medication drops and, ultimately, surgery. The type of surgery is decided by determining the severity and progress of an individual's vision loss.

Certain glaucoma surgeries (including PreserFlo microshunts, and Xen stents) involve creation of an alternative passage for the liquid inside of the eye to be drained. Glaucoma surgery is complex and excessive inflammation and scarring can increase pressure inside the eye and lead to surgical failure. We hope that covering PreserFlo microshunts and Xen stents with amniotic membrane will result in reduced scarring and better pressure outcomes after these surgeries.

Previous research has shown that amniotic membrane is safe for the eye and has improved the outcomes of other similar glaucoma surgeries. However, there are no studies that have investigated whether amniotic membrane is a safe and effective in PreserFlo microshunts, and Xen stents surgeries.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and older
2. Patients selected for PreserFlo microshunt surgery and XEN stent alone or in combination with cataract surgery.
3. Ability to comprehend the study procedures

Exclusion Criteria:

1. Unwilling or unable to give consent
2. Unable to come for scheduled post-operative visits
3. Pregnant or nursing women
4. Previous cyclodestructive procedures, scleral buckling procedures, or presence of silicone oil
5. Conjunctival scarring precluding a glaucoma surgery superiorly
6. Active iris neovascularization or active proliferative retinopathy
7. Vitreous in the anterior chamber for which a vitrectomy is anticipated.
8. Previous trabeculectomy, tube-shunt implantation, or surgeries that shunt aqueous outflow into the subconjunctival space

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of adverse events | Surgery (Day 0) to 12 months
  Proportion of study eyes with ≥1 of: persistent uveitis, blebitis, endophthalmitis, clinically significant hypotony, stent erosion, bleb dysesthesia, or loss of best-corrected visual acuity. Each AE recorded as yes/no; between-group comparisons via logistic regression (adjusting for device type and baseline IOP).
Relative Reduction in Intraocular Pressure (IOP) at 3, 6, and 12 Months | Baseline to 3, 6, and 12 months
  Percent change from baseline IOP at each post-operative visit. Calculated per study eye as:
  [(Baseline IOP - Visit IOP) / Baseline IOP] × 100. Primary efficacy analysis uses a linear mixed-effects model (repeated measures) with fixed effects for treatment group (amniotic membrane vs no membrane), visit (3/6/12 months), treatment × visit interaction, device type (PreserFlo vs XEN), and baseline IOP; participant (study eye) included as a random effect. Estimates will report least-squares mean differences between groups in percent reduction at each visit and an overall treatment effect across visits, with 95% confidence intervals and p-values

SECONDARY OUTCOMES:
Number of re-operations | Through 12 months post-op
  To compare the number of re-operations per patient at 12 months between the treatment groups, we will use a negative binomial regression model. The dependent variable will be the total number of re-operations per patient, and the independent variable will be the treatment group. Results will be reported as incidence rate ratios (IRRs) with 95% confidence intervals and p-values.
Number of Glaucoma Medications | 3, 6 and 12 month post-op
  Count of post-operative glaucoma medication classes required at each visit. Generalized linear mixed model with negative binomial distribution compares groups over time; reported as rate ratios with 95% CIs and p-values.
Time to Surgical Failure | From surgery to 12 months post-op (failures assessed after postoperative Month 3)
  Failure is defined as any of: (a) IOP >21 mmHg or <20% reduction from baseline on two consecutive visits; (b) IOP ≤5 mmHg on two consecutive visits (hypotony); (c) any re-operation for glaucoma; or (d) loss of light perception vision. Analyzed by Kaplan-Meier and Cox proportional hazards; reported as hazard ratio with 95% CI and p-value.